CLINICAL TRIAL: NCT06760637
Title: AN INTERVENTIONAL, OPEN-LABEL, RANDOMIZED, MULTICENTER PHASE 3 STUDY OF PF-07220060 PLUS LETROZOLE COMPARED TO CDK4/6 INHIBITOR PLUS LETROZOLE IN PARTICIPANTS OVER 18 YEARS OF AGE WITH HORMONE RECEPTOR (HR)-POSITIVE, HER2-NEGATIVE ADVANCED/METASTATIC BREAST CANCER WHO HAVE NOT RECEIVED ANY PRIOR SYSTEMIC ANTICANCER TREATMENT FOR ADVANCED/METASTATIC DISEASE (FOURLIGHT-3)
Brief Title: Study of PF-07220060 With Letrozole in Adults With HR-positive HER2-negative Breast Cancer Who Have Not Received Anticancer Treatment for Advanced/Metastatic Disease
Acronym: FourLight-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C4391024; 2024-512925-95-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2024-12-11; First posted 2025-01-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: Locally advanced or metastatic breast cancer; Estrogen receptor positive [ER(+)]; Progesterone receptor positive [PR(+)]; Hormone receptor positive [HR(+)]; Human epidermal growth factor receptor 2 negative [HER2(-)]; ER(+)/HER2(-); PR(+)/HER2(-); HR(+)/HER2(-); Advanced Breast Cancer; Breast tumor; Breast cancer; Palbociclib; Abemaciclib; Ribociclib; Partial Response+ (PR+); Metastatic breast cancer; Hormone Therapy; Hormone positive breast cancer; Recurrent breast cancer; HR+; HER2-negative; Relapse; Recurrent; First line treatment; Left Sided Breast Cancer; Left-Sided Breast Cancer; Right Sided Breast Cancer; Right-Sided Breast Cancer; Unilateral Breast Cancer; Cancer of the breast; CDK4i; CDK4/6i; Bilateral Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Recurrence; Unilateral Breast Neoplasms | interventions — Letrozole; abemaciclib; palbociclib; ribociclib

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned into 1 of 2 groups in parallel for the entire duration of the study. The experimental arm will receive PF-07220060 and letrozole (Arm A) while the comparator arm with receive the study doctors choice of CDK4/6i and letrozole (Arm B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): PF-07220060 tablet taken by mouth plus Letrozole tablet taken by mouth
  Interventions: Drug: PF-07220060; Drug: letrozole
- Arm B (Active Comparator): Investigator's Choice of CDK4/6 inhibitor (tablet/capsule) taken by mouth with letrozole tablet taken by mouth
  Interventions: Drug: letrozole; Drug: abemaciclib; Drug: palbociclib; Drug: ribociclib

INTERVENTIONS:
Drug: PF-07220060 — CDK4 inhibitor
  Arms: Arm A
Drug: letrozole — endocrine therapy
Drug: abemaciclib — CDK4/6 inhibitor
  Arms: Arm B
Drug: palbociclib — CDK4/6 inhibitor
  Arms: Arm B
Drug: ribociclib — CDK4/6 inhibitor
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine the safety and efficacy of PF-07220060 with letrozole compared to approved treatments (ie, palbociclib, ribociclib or abemaciclib with letrozole) in people with breast cancer:

* HR-positive (breast cancer cells that need estrogen or progesterone to grow)
* HER2-negative (cells that have a small amount or none of a protein called HER2 on their surface);
* locally advanced (that has spread from where it started to nearby tissue or lymph nodes) or metastatic disease (the spread of cancer to other places in the body)
* who have not received any prior systemic anti-cancer treatment for advanced/metastatic disease.

Approximately half of the participants will receive PF-07220060 plus letrozole while the other half of participants will receive the investigator's choice of treatment plus letrozole.

The study team will monitor how each participant is doing with the study treatment during regular visits at the study clinic.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of breast cancer with evidence of locally advanced or metastatic disease, which is not amenable to surgical resection or radiation therapy with curative intent.
* Documented estrogen receptor (ER) and/or progesterone receptor (PR)-positive tumor
* Documented HER2-negative tumor
* Previously untreated with any systemic anticancer therapy for their locally advanced or metastatic disease.
* Measurable disease or non-measurable bone only disease as defined by RECIST version 1.1

Exclusion Criteria:

* In visceral crisis at risk of immediately life-threatening complications in the short term.
* Current or past history of central nervous system metastases.
* Have received prior (neo)adjuvant endocrine therapy (ET) and had recurrence during or within 12 months after the last dose of ET.
* Have received prior (neo)adjuvant CDK4/6i and had recurrence during or within 12 months after the last dose of CDK4/6i.
* Inadequate renal function, hepatic dysfunction, or hematologic abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2037-12-29 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) by BICR | From the date of randomization until disease progression or death due to any cause (up to approximately 4 years)
  Time from the date of randomization to the date of the first documentation of objective progressive disease as determined by blinded independent central review (BICR) per RECIST v1.1, or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of randomization until death due to any cause (up to approximately 13 years).
  Time from the date of randomization to the date of death due to any cause
Progression Free Survival (PFS) by Investigator | From the date of randomization until disease progression or death due to any cause (up to approximately 4 years)
  Time from the date of randomization to the date of the first documentation of objective progressive disease as determined by investigator per RECIST v1.1, or death due to any cause, whichever occurs first
OR by BICR and by investigator | From randomization to progression or death whichever occurs first (up to approximately 4 years)
  Time from randomization date (every 8 weeks during the first 48 weeks and then every 12 weeks) to the date of progression OR death whichever occurs first
Duration of Response (DoR) by BICR and by investigator | From the date of CR or PR until objective progressive disease, or death (up to approximately 4 years)
  Time from the date of CR or PR to the first documentation of objective progressive disease, or death due to any cause, whichever occurs first
Incidence of treatment emergent treatment related adverse events (AE) | Duration of the study approximately up to 13 years.
  Incidence and severity of AEs graded according to the NCI CTCAE v5.0
Incidence of treatment emergent treatment related serious adverse events | Duration of the study approximately up to 13 years.
  Incidence and severity of AEs graded according to NCI CTCAE v5.0
Estimated mean change from baseline in EORTC QLQ C30 | Baseline to end of treatment (up to approximately 4 years)
Estimated mean change from baseline in BPI-SF | Baseline to end of treatment (up to approximately 4 years)
Estimated mean change from baseline in EQ-5D-5L | Baseline to end of treatment (up to approximately 4 years)
Estimated mean change from baseline in EORTC Breast Cancer Module (BR42) | Baseline to end of treatment (up to approximately 4 years)
Mean change from baseline of ctDNA | Baseline to end of treatment (up to approximately 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (449):
- United States (170):
  - The Kirklin Clinic of UAB Hospital, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Ironwood Cancer & Research Centers, Gilbert, Arizona
  - Ironwood Cancer & Research Centers, Glendale, Arizona
  - Ironwood Cancer & Research Centers, Goodyear, Arizona
  - Ironwood Cancer & Research Centers, Mesa, Arizona
  - Ironwood Cancer & Research Centers, Phoenix, Arizona
  - Ironwood Cancer & Research Centers, Scottsdale, Arizona
  - CARTI Cancer Center Saline County, Bryant, Arkansas
  - CARTI Cancer Center Conway, Conway, Arkansas
  - Highlands Oncology, Fayetteville, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - CARTI Cancer Center North Little Rock Urology, North Little Rock, Arkansas
  - CARTI Cancer Center North Little Rock, North Little Rock, Arkansas
  - CARTI Cancer Center Pine Bluff, Pine Bluff, Arkansas
  - Highlands Oncology, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Cedars-Sinai Cancer Beverly Hills (drug treatment and dispensing location), Beverly Hills, California
  - Cedars-Sinai Cancer Beverly Hills, Beverly Hills, California
  - Premier Cancer Care and Infusion Center - Fresno - North Thesta Street, Fresno, California
  - Providence Medical Foundation, Fullerton, California
  - Providence St. Jude Medical Center, Fullerton, California
  - Cancer and Blood Research Center, LLC, Los Alamitos, California
  - Cancer and Blood Specialty Clinic / Cancer and Blood Research Center, LLC, Los Alamitos, California
  - San Vicente Surgical Center, Los Angeles, California
  - Keck Hospital of USC, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - Norris Healthcare Center 3 (HC3), Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars-Sinai Cancer at Cedars-Sinai Medical Center (drug treatment and dispensing location), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Keck Medicine of USC Norris Oncology/Hematology - Newport Beach Treatment Center, Newport Beach, California
  - USC Norris Oncology/Hematology - Newport Beach, Newport Beach, California
  - Clinical and Translational Research Unit (CTRU), Palo Alto, California
  - Stanford Cancer Center, Palo Alto, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Health - Sutter Institute for Medical Research, Sacramento, California
  - Stanford Health Care, Investigational Drug Service, Stanford, California
  - Cancer AND Blood Specialty Clinic, Torrance, California
  - Hunt Cancer Institute, an Affiliate of Cedars-Sinai Cancer, Torrance, California
  - Wellness Oncology Hematology, West Hills, California
  - Breast Health Services Building, West Hollywood, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - Intermountain Health St. Joseph Hospital, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Intermountain Health Lutheran Hospital, Golden, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - Cancer Centers of Colorado St. Mary's Regional Hospital, Grand Junction, Colorado
  - Intermountain Health Saint Mary's Regional Hospital, Grand Junction, Colorado
  - Intermountain Health, Grand Junction, Colorado
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte Infusion Center, Altamonte Springs, Florida
  - AdventHealth Altamonte Springs, Altamonte Springs, Florida
  - AdventHealth Medical Group Altamonte, Altamonte Springs, Florida
  - Mount Sinai Medical Center, Aventura, Aventura, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - AdventHealth Orlando, Orlando, Florida
  - AdventHealth Medical Group Orlando, Orlando, Florida
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - Grady Health System Correll Pavilion, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Emory Johns Creek Hospital, Johns Creek, Georgia
  - Summit Cancer Care, PC, Savannah, Georgia
  - St. Luke's Cancer Institute: Boise, Boise, Idaho
  - St. Luke's Regional Medical Center, Boise, Idaho
  - St. Luke's Cancer Institute-Fruitland, Fruitland, Idaho
  - St. Luke's Cancer Institute-Meridian, Meridian, Idaho
  - St. Lukes Meridian Medical Center, Meridian, Idaho
  - St. Luke's Cancer Institute-Nampa, Nampa, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - AMG Crystal Lake -Oncology, Crystal Lake, Illinois
  - Endeavor Health, Elmhurst, Illinois
  - Prime Saint Francis-Infusion Services Evanston, Evanston, Illinois
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - AMG - Libertyville, Libertyville, Illinois
  - Endeavor Health, Naperville, Illinois
  - Hope and Healing Cancer Services, New Lenox, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Advocate Medical Group, Park Ridge, Illinois
  - Memorial Hospital, Shiloh, Illinois
  - Siteman Cancer Center - Shiloh, Shiloh, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Prime Saint Francis-Infusion Services Skokie, Skokie, Illinois
  - Velocity Clinical Research, Annapolis, Maryland
  - Mercy Medical Center - Baltimore, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center (Investigational Pharmacy services, IP delivery), Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Chestnut Hill, Newton, Massachusetts
  - Allina Health Cancer Institute - Mercy Hospital, Coon Rapids, Minnesota
  - Allina Health Cancer Institute - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Allina Health Cancer Institute - United Hospital, Saint Paul, Minnesota
  - Siteman Cancer Center - St Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Siteman Cancer Center - North County, Florissant, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Renown Health Medical Oncology, Reno, Nevada
  - Renown Office of Clinical Research, Reno, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Renown Health Conrad Breast Center, Reno, Nevada
  - Renown Research Office - South Meadows, Reno, Nevada
  - Renown South Meadows Medical Center, Reno, Nevada
  - Jersey City Medical Center, Jersey City, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Stony Brook University, Stony Brook, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - University of North Carolina Hospitals at Hillsborough, Hillsborough, North Carolina
  - Oncology Associates of Oregon, P.C., Albany, Oregon
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center Investigational Drug Services, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Investigational Drug Service - Westside, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic - Westside, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Oncology Associates of Oregon, P.C., Springfield, Oregon
  - US Oncology Investigational Products Center, Irving, Texas
  - US Oncology lnvestigational Products Center (IPC), Irving, Texas
  - Baylor Scott & White Medical Center - Round Rock, Round Rock, Texas
  - The University of Texas Health Science Center at Tyler dba UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - The University of Texas Health Science Center at Tyler on behalf of UT Health East Texas HOPE Cancer, Tyler, Texas
  - Utah Cancer Specialists, Bountiful, Utah
  - Utah Cancer Specialists, Layton, Utah
  - Utah Cancer Specialists, Murray, Utah
  - Utah Cancer Specialists, Ogden, Utah
  - Utah Cancer Specialists, Orem, Utah
  - Utah Cancer Specialists, Pleasant Grove, Utah
  - Utah Cancer Specialists, Provo, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Utah Cancer Specialists, West Jordan, Utah
  - Utah Cancer Specialists, West Valley City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Manassas, Virginia
  - Bon Secours Cancer Institute at Memorial Regional, Mechanicsville, Virginia
  - Bon Secours St. Francis Medical Center, Midlothian, Virginia
  - Virginia Cancer Specialists, PC, Reston, Virginia
  - Bon Secours Cancer Institute at St. Mary's, Richmond, Virginia
  - Aurora Medical Center, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Cancer Care - Milwaukee / Good Hope, Milwaukee, Wisconsin
  - Aurora Cancer Care, Milwaukee, Wisconsin
  - Aurora St Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
- Argentina (4):
  - Organizacion Medica de Investigacion, CABA, Buenos Aires
  - CIPREC, Buenos Aires, Buenos Aires F.D.
  - Fundación Respirar, Buenos Aires
  - Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
- Australia (6):
  - Townsville University Hospital, Douglas, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Rosebud Hospital, Capel Sound, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Belgium (5):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Grand Hôpital de Charleroi, Gilly, Hainaut
  - AZ Maria Middelares, Ghent, Oost-vlaanderen
  - UZ Leuven, Leuven, Vlaams-brabant
  - AZORG Campus Aalst-Moorselbaan, Aalst
- Brazil (6):
  - Hospital Brasilia, Brasília, Federal District
  - Santa Casa de Misericordia de Passos, Passos, Minas Gerais
  - Associação Hospitalar Beneficente São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Icesp - Instituto Do Câncer Do Estado de São Paulo, São Paulo
- Bulgaria (8):
  - Multiprofile Hospital for Active Treatment Serdikamed EOOD, Sofia, Sofia (stolitsa)
  - Complex Oncology Center - Burgas, Burgas
  - Multiprofile Hospital for Active Treatment Dr. Tota Venkova AD, Gabrovo
  - Specialized Hospital for Active Treatment of Oncology - Haskovo, Haskovo
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Complex Oncology Center - Shumen, Shumen
  - MHAT for Women's Health Nadezhda, Sofia
  - University Specialized Hospital for Active Treatment of Oncology EAD, Sofia
- Canada (6):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Dr. Everett Chalmers Regional Hospital, Fredericton, New Brunswick
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- China (29):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Wuhan Union Hospital Cancer Center, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Nanchang People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The 2nd Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Czechia (6):
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Fakultni nemocnice v Motole, Prague, Praha 5
  - Fakultni nemocnice Bulovka, Prague, Praha 8
  - Nemocnice AGEL Novy Jicin a.s., Nový Jičín
  - Fakultni nemocnice Kralovske Vinohrady, Prague
- Denmark (8):
  - Rigshospitalet, Copenhagen, Capital Region
  - Herlev and Gentofte Hospital, Copenhagen, Capital Region
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
  - Aalborg Universitetshospital, Syd, Aalborg, North Denmark
  - Næstved Sygehus, Næstved, Region Sjælland
  - Esbjerg sygehus, Syddansk Universitetshospital, Esbjerg, Region Syddanmark
  - Odense Universitetshospital, Odense, Region Syddanmark
  - Sygehus Soenderjylland, Sønderborg, Region Syddanmark
- Finland (5):
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Vaasan Keskussairaala, Vaasa, Pohjanmaa
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University Hospital - Comprehensive Cancer Center (HYKS - Syöpäkeskus), Helsinki, Uusimaa
  - Satakunnan Keskussairaala, Pori
- France (12):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux, Aquitaine
  - Centre Oscar Lambret, Lille, Hauts-de-France
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer, Rennes, Ille-et-vilaine
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-roussillon
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-atlantique
  - Institut de Cancérologie de l'Ouest, Angers, Maine-et-loire
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen, Rouen, Seine-maritime
  - Gustave Roussy, Villejuif, Val-de-marne
  - CHD Vendee, La Roche-sur-Yon, Vendée
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Henri Mondor Hospital, Créteil, Île-de-France Region
- Germany (7):
  - MVZ für Hämatologie und Onkologie Ravensburg GmbH - Studienzentrum, Ravensburg, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - InVO Institut für Versorgungsforschung in der Onkologie, Koblenz, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden, Saxony
  - Gemeinschaftspraxis Hämatologie - Onkologie Freiberg-Richter, Jacobasch, Illmer, Wolf, Dresden
  - Facharztzentrum Eppendorf, Hamburg
  - MVZ für Hämatologie und Onkologie, Velbert
- Greece (6):
  - Agios Savvas Regional Cancer Hospital, Athens, Attikí
  - Aretaieio Hospital, Athens, Attikí
  - Hygeia Hospital, Marousi, Attikí
  - University General Hospital of Heraklion, Heraklion, Irakleío
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki, Thessaloníki
  - Aretaieio Hospital, Athens
- Hungary (5):
  - Borsod-Abaúj-Zemplén Vármegyei Központi Kórház és Egyetemi Oktatókórház, Miskolc, Borsod-Abauj Zemplen county
  - Heves Vármegyei Markhot Ferenc Oktatókórház és Rendelőintézet, Eger, Heves County
  - Szabolcs Szatmár Bereg Vármegyei Oktatókórház, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Országos Onkológiai Intézet, Budapest
  - Budapesti Uzsoki Utcai Kórház, Budapest
- India (11):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - Artemis hospital, Gurugram, Haryana
  - Spandana Oncology Centre (SOC), Bangalore, Karnataka
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - Apex Wellness Hospital, Nashik, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - Bhakti Vedanta Hospital and Research Institute, Thane, Maharashtra
  - Rajiv Gandhi Cancer Institute And Research Centre, New Delhi, National Capital Territory of Delhi
  - Basavatarakam Indo American Cancer Hospital & Research Institute, Hyderabad, Telangana
  - Apollo Multispeciality Hospitals limited, Kolkata, West Bengal
- Ireland (5):
  - St. Vincent's University Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - Mater Private Hospital - Dublin, Dublin
  - St. James's Hospital, Dublin
  - Beaumont Hospital, Dublin, Dublin
- Israel (5):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Northern District
  - Sourasky Medical Center, Tel Aviv, TELL ABĪB
- Italy (11):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, Emilia-Romagna
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Cro-Irccs, Aviano, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Rome, Lazio
  - Istituto Nazionale Tumori Regina Elena, Rome, ROMA
  - Ospedale Isola Tiberina - Gemelli Isola, Rome, ROMA
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero Universitaria Maggiore della Carità, Novara
  - Istituto Oncologico Veneto IRCCS, Padua
- Japan (21):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Gunma Prefectural Cancer Center, Otashi, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa cancer center, Yokohama, Kanagawa
  - Kyoto University Hospital, Sakyo-ku, Kyoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka University Hospital, Suita, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Showa University Hospital, Shinagawa, Tokyo
  - National Center for Global Health and Medicine, Shinjuku, Tokyo
  - Chiba Cancer Center, Chiba
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Kumamoto Shinto General Hospital, Kumamoto
  - Okayama University Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
- Mexico (4):
  - Boca Clinical Trials Mexico S.C., Guadajalara, Jalisco
  - COI Centro Oncologico Internacional S.A.P.I. de C.V., Mexico City, Mexico City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - Instituto Veracruzano en Investigación Clínica S.C., Veracruz
- Netherlands (6):
  - VieCuri Medisch Centrum, locatie Venlo, Venlo, Limburg
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Amphia Ziekenhuis, locatie Breda Molengracht, Breda, North Brabant
  - Spaarne Gasthuis - Hoofddorp, Hoofddorp, North Holland
  - Frisius Medisch Centrum, Leeuwarden, Provincie Friesland
  - Meander Medisch Centrum, Amersfoort, Utrecht
- Poland (10):
  - AIDPORT Sp. z o.o., Skórzewo, Greater Poland Voivodeship
  - Regionalny Szpital Specjalistyczny im. dr. Władyslawa Biegańskiego, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Centrum Badań Klinicznych Jagiellońskie Centrum Innowacji sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - WSD MEDI, Warsaw, Masovian Voivodeship
  - Białostockie Centrum Onkologii im. M. Skłodowskiej-Curie w Białymstoku, Bialystok, Podlaskie Voivodeship
  - Szpitale Pomorskie Sp. z o. o., Gdynia, Pomeranian Voivodeship
  - Szpital Wojewódzki im. Mikoaja Kopernika w Koszalinie, Koszalin, West Pomeranian Voivodeship
  - Europejskie Centrum Zdrowia Otwock Szpital im.F.Chopina, Otwock
  - Instytut MSF Sp zoo, Lodz, Łódź Voivodeship
- Slovakia (6):
  - Narodny onkologicky ustav, Bratislava, Bratislava Region
  - Nemocnica s poliklinikou Stefana Kukuru Michalovce a.s., Michalovce, Košice Region
  - Nemocnica AGEL Komarno, Komárno, Nitra Region
  - Medeon, s.r.o., Banka, Trnava Region
  - Fakultna nemocnica Trnava, Trnava, Trnava Region
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky
- South Korea (14):
  - Gachon University Gil Medical Center, Incheon, Incheon-gwangyeoksi [incheon]
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Kyǒnggi-do
  - Gangnam Severance Hospital, Yonsei University Health System, Gangnam-gu, Seoul-teukbyeolsi [seoul]
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Kangbuk Samsung Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (20):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [LA Coruña]
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, Hospitalet, Barcelona [barcelona]
  - Osi Bilbao-Basurto, Bilbao, Basque Country
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia, Región de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Fundación Instituto Valenciano de Oncología, Valencia, Valenciana, Comunitat
  - Hospital Arnau de Vilanova, Valencia, València
  - Hospital Universitario San Cecilio, Granada
  - Hospital Beata María Ana, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
- Sweden (9):
  - Sjukhuset I Gävle, Gävle, Gävleborgs LÄN [se-21]
  - Karolinska Universitetssjukhuset Solna, Solna, Stockholms LÄN [se-01]
  - Södersjukhuset, Stockholm, Stockholms LÄN [se-01]
  - Akademiska sjukhuset, Uppsala, Uppsala LÄN [se-03]
  - Västmanlands Sjukhus Västerås, Västerås, Västmanlands LÄN [se-19]
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands LÄN [se-14]
  - Lanssjukhuset Ryhov, Jönköping
  - Capio Saint Görans Sjukhus, Stockholm
  - Sundsvalls Sjukhus, Sundsvall
- Switzerland (11):
  - Tumor Zentrum Aarau, Aarau, Canton of Aargau
  - University Hospital Basel, Basel, Canton of Basel-City
  - Inselspital Bern, Bern, Canton of Bern
  - CHUV (centre hospitalier universitaire vaudois), Lausanne, Canton of Vaud
  - Kantonsspital Frauenfeld - Spital Thurgau AG, Frauenfeld, Thurgau
  - UniversitätsSpital Zürich, Zurich, Zürich (DE)
  - Kantonsspital Baden, Baden
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Münsterlingen - Spital Thurgau AG, Münsterlingen
  - Kantonsspital Olten, Olten
  - Kantonsspital Winterthur, Winterthur
- Taiwan (8):
  - National Taiwan University Hospital - Hsinchu branch, Zhubei, Hsinchu
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (13):
  - Medipol Mega Universite Hastanesi, Istanbul, İ̇stanbul
  - İ.A.Ü VM Medical Park Florya Hastanesi, Istanbul, İ̇stanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul, İ̇stanbul
  - Ege Universitesi Hastanesi, Izmir, İ̇zmir
  - Adana Medical Park Seyhan Hastanesi, Adana
  - Adana City Hospital, Adana
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastırma Hastanesi, Ankara
  - Hacettepe Universite Hastaneleri, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Gazi University Health Research and Application Center Gazi Hospital, Ankara
  - Dicle Üniversitesi, Diyarbakır
  - Sakarya Training and Research Hospital, Sakarya
- United Kingdom (12):
  - Derriford Hospital, Plymouth, Devon
  - The Princess Alexandra Hospital NHS Trust, Harlow, England
  - The Royal Cornwall Hospital, Truro, England
  - Imperial College Healthcare NHS Trust, Charing Cross Hospital, London, Hammersmith and Fulham
  - Maidstone Hospital, Maidstone, KENT
  - Sarah Cannon Research Institute UK, London, London, CITY of
  - Western General Hospital, Edinburgh, Midlothian
  - Musgrove Park Hospital, Taunton, Somerset
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - University Hospital Coventry & Warwickshire, Coventry, Warwickshire
  - Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391024